CLINICAL TRIAL: NCT02314325
Title: Subclinical Joint Bleeding in Irish Adults With Severe Haemophilia A on Personalised Prophylaxis Regimens
Acronym: PERSONAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Collaborators: Baxter BioScience (Industry)
Responsible Party: Principal Investigator, Dr. Niamh O'Connell, Consultant Haematologist, St. James's Hospital, Ireland
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-003240-23
Record Dates: First submitted 2014-09-03; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Severe Haemophilia A
Keywords: Factor VIII deficiency; Arthropathy; MRI; XRay; Joint; HJHS
MeSH Terms: conditions — Hemophilia A; Joint Diseases | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard prophylaxis (Active Comparator): Advate [Antihemophilic Factor(Recombinant)] 20-40 IU/kg 5-7 infusions per 14days
  Interventions: Drug: ADVATE [Antihemophilic Factor (Recombinant)]
- Pharmacokinetic tailored prophylaxis (Experimental): Advate [Antihemophilic Factor(Recombinant)] dose determined by individual patient pharmacokinetics and infusions administerd on alternate days
  Interventions: Drug: ADVATE [Antihemophilic Factor (Recombinant)]

INTERVENTIONS:
Drug: ADVATE [Antihemophilic Factor (Recombinant)] — In Arm 1 prior patients will be dosed as per body weight 20-40 IU/kg 5-7 infusions per fortnight
  Arms: Standard prophylaxis
Drug: ADVATE [Antihemophilic Factor (Recombinant)] — In Arm 2 patients who have completed arm 1 will cross over onto an individualised PK tailored alternate day dosing regimen
  Arms: Pharmacokinetic tailored prophylaxis

SUMMARY:
This trial is designed to assess if there is evidence of subclinical joint bleeding on MRI/X-Ray in adults with severe Haemophilia A while on standard and/or pharmacokinetically tailored prophylaxis regimens. Participants with severe Haemophilia A will have longitudinal MRI and XRay imaging of their elbows, ankles and knees at 0, 6 and 18 months while on standard ( 0-6 months) and then pharmacokinetically tailored (7-18 months) recombinant Factor VIII prophylaxis.

DETAILED DESCRIPTION:
Subclinical joint bleeding (SJB) in Haemophilia may cause early and progressive joint damage. Clinical haemarthrosis is a traditional outcome measure in Haemophilia trials but may not always correlate with the degree of arthropathy. Even in the absence of haemarthrosis, abnormalities may be detected on MRI. MRI offers greater sensitivity than physical examination for early joint damage and use of the International Prophylaxis Study Group (IPSG) score allows standardisation across clinical trials. Early awareness of haemophiliac arthropathy can prompt intervention with physiotherapy, specific exercise programmes, optimization of prophylaxis and orthotics to improve overall joint outcomes.

The time spent with Factor VIII (FVIII) levels <0.01 IU/mL is a known risk for bleeding. Conventional prophylaxis schedules follow a weight based regimen and are titrated according to clinical bleeds. FVIII pharmacokinetics (PK) may be used to optimise FVIII prophylactic regimens, maintaining adequate FVIII trough levels. This offers the possibility to not only tailor individual regimens but also may potentially reduce the rate of clinical and subclinical joint bleeding.

This is a national, investigator led clinical trial investigating the feasibility of PK tailored prophylaxis in adults with severe Haemophilia A. This trial will prospectively and longitudinally assess SJB and joint health in Irish adults with severe Haemophilia A.

SJB will be compared while on standard (weight based, 20-40 IU/kg) and PK tailored prophylaxis(maintaining trough FVIII > 0.015 IU/mL). This is a crossover study will participants spending months 0-6 on standard prophylaxis and then changing over to PK tailored dosing for months 7-18. A comprehensive joint assessment involving bleed history, clinical examination, physical activity, specialist physiotherapy review, X-rays and MRI scanning of bilateral ankles, knees and elbow will be performed at months 0,6 and 18. Haemophilia Joint Health Score (HJHS), International Physical Activity (IPAQ) and EuroQoL 5-Dimensions (EQ5D) Questionnaires will also be performed at these three timepoints.

Clinical bleeds and FVIII usage will be recorded throughout the trial using the investigators Home Scan system, a smart phone application that allows patients to log factor VIII usage.

Results will be compared between both arms and between participants on primary and secondary prophylaxis. Information on those with naïve joints versus established arthropathy will be compared.

Due to the relative rarity of severe Haemophilia A the investigators plan to recruit 20 patients in total. All patients will act as their own control, crossing over from standard to PK tailored prophylaxis with joint assessments prior to crossover to allow comparison of the two regimes.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with severe Haemophilia A (baseline Factor VIII level of <0.01 IU/mL)
* Age 18 years and above
* Patients taking any regular prophylactic regimen (defined as regular factor VIII infusions, at least 5 times a fortnight, with the aim of minimising haemarthroses and other clinically significant bleeds).
* Low titre inhibitors, past history of an inhibitor, abnormal liver function, drugs that interfere with haemostasis and low Cluster of Differentiation 4 (CD4) counts are allowed.

Exclusion Criteria:

* Presence of a target joint on prophylaxis (defined as 3 bleeds into one joint, during a 6 month period, during the last year).
* The occurrence of more than 3 haemarthroses in the last year that required more than 2 infusions to resolve.
* Patients with a learning disability or dementia
* Prisoners
* Adults who are unconscious/unable to give informed consent
* Participants with a pacemaker or implanted medical devices which are unsuitable to have a MRI will be excluded from the MRI scans during the trial but may proceed with other components.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Number of subclinical haemarthroses | 18 months
  The number of subclinical haemarthroses identifed on serial MRI scans of elbow, knee and ankle joints

SECONDARY OUTCOMES:
EQ5D QoL score | 18 months
  Comparison of score on EQ5D Quality of life questionnaire on standard versus PK tailored dosing
Percentage of prescribed doses of prophylaxis taken | 18 months
  The number of missed doses of prophylaxis on the standard and PK tailored dosing regimens
IPAQ score | 18 months
  Comparison of IPAQ activity scores (numeric) on standard versus PK tailored dosing
Haemophilia joint health score (HJHS) | 18 months
  Comparison of HJHS numeric score on standard versus PK tailored dosing
Amount of FVIII usage (units) | 18 months
  Comparison of FVIII usage in units on standard versus PK tailored dosing
MRI joint score | 18 months
  Comparison of joint score (numeric) determined on MRI by the International prophylaxis study group (IPSG) score
Petterson joint score | 18 months
  Comparison of Petterson joint score (numeric) on plain films for patients on standard versus PK tailored dosing
Number of clinical haemarthroses | 18 months
  Number of patient reported haemarthroses on standard prophylaxis versus PK tailored prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Niamh M O'Connell, PhD, FRCPath, Principal Investigator — St. James's Hospital, Ireland; James O'Donnell, PhD, FRCPath, Principal Investigator — St. James's Hospital, Ireland
Locations (1):
- St. James's Hospital, Dublin, Dublin, Ireland